CLINICAL TRIAL: NCT04799093
Title: Eye Movement Tracking to Detect Impairment Due to Acute Cannabis Intoxication
Status: Completed | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-B
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Impairment; Cannabis Intoxication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cannabis users
  Interventions: Diagnostic Test: EyeBOX
- Normals
  Interventions: Diagnostic Test: EyeBOX

INTERVENTIONS:
Diagnostic Test: EyeBOX — Eye-Tracking based diagnostic

SUMMARY:
The purpose of this study is to determine the accuracy of an impairment algorithm based on eye tracking while watching a short film clip, in comparison to a clinical reference standard of impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Have the ability to provide a complete ophthalmologic, medical and neurologic history as well as report medications/drugs/alcohol consumed within the 24 hours prior to tracking.
3. Be at least 18 years old.

Exclusion Criteria:

1. Be blind (no light perception), have missing or non-functional eyes.
2. Be unable to open their eyes.
3. Have a history of unresolved strabismus, diplopia, amblyopia.
4. Have a history of unresolved cranial nerve III, IV, or VI palsy.
5. Have a history of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption.
6. Have a history of extensive prior eye surgery (examples include strabismus surgery, scleral buckle repair of retinal detachment, repair of blow out fractures of the orbit and any procedures that would interfere with extraocular muscle movements; prior cataract surgery or Lasik are not exclusions) or scarring.
7. Have a prior history of unresolved ocular-motor dysfunctions.
8. Have used cannabis, alcohol etc. 24 hours before study commences.
9. Be 100% naïve to cannabis usage.
10. Be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy habitual cannabis-smoking subjects, i.e., smoke or consume cannabis at least three times a week, and healthy occasional cannabis-smoking subjects, i.e., smoke or consume once a week will be recruited from the local area.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Impairment assessment correlation with EyeBOX assessment | Within an hour
  A correlation between impairment as assessed by standard impairment tests and the EyeBOX assessment of impairment as determined by an algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Rosina Samadani, Ph.D., Study Director — Oculogica, Inc.
Locations (1):
- Integrated Medicine LLC, Westport, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No